CLINICAL TRIAL: NCT02066922
Title: A Comparative Study of Two Daily Disposable Contact Lenses in Higher Myopia Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: C-12-057
Record Dates: First submitted 2013-08-08; First posted 2014-02-20 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Refractive Error; Myopia
Keywords: Contact lenses; Nearsightedness; Corneal curvature; K-reading; High minus; Spectacle refraction
MeSH Terms: conditions — Refractive Errors; Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAILIES TOTAL1 (Experimental): Delefilcon A contact lens randomly assigned to one eye, with narafilcon A contact lens in the fellow eye for contralateral wear. Both products worn in a daily wear, daily disposable mode approximately 8 hours a day for approximately 1 week, with spectacles worn over contact lenses if needed to provide acceptable vision.
  Interventions: Device: Delefilcon A contact lens; Device: Narafilcon A contact lens; Device: Spectacles
- TRUEYE (Active Comparator): Narafilcon A contact lens randomly assigned to one eye, with delefilcon A contact lens in the fellow eye for contralateral wear. Both products worn in a daily wear, daily disposable mode approximately 8 hours a day for approximately 1 week, with spectacles worn over contact lenses if needed to provide acceptable vision.
  Interventions: Device: Delefilcon A contact lens; Device: Narafilcon A contact lens; Device: Spectacles

INTERVENTIONS:
Device: Delefilcon A contact lens — Commercially available silicone hydrogel contact lens
  Other Names: DAILIES® TOTAL1®
Device: Narafilcon A contact lens — Commercially available silicone hydrogel contact lens
  Other Names: 1-DAY ACUVUE TRUEYE™
Device: Spectacles — Incremental prescription worn over contact lenses if needed to provide acceptable vision

SUMMARY:
The purpose of this study is to compare the change from baseline in central corneal curvature at one week, between 2 silicone hydrogel lenses, in higher myopic subjects.

DETAILED DESCRIPTION:
Participants were expected to attend 4 office visits. Visit 1 was the Screening/Enrollment visit. At Visit 2 (Baseline Visit), participants were randomized and the study lenses were trial fit. At Visit 3 (Dispense Visit), participants received study lenses for approximately 1 week of wear. Visit 4 was the Exit visit. Expected duration of participation in the study was 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent document;
* Higher degree of myopia in both eyes, i.e. habitual contact lens power between -10.00 diopters (D) and -17.00D;
* Best corrected distance visual acuity greater than or equal to 20/30 in each eye (measured with either spectacle refraction or habitual contact lenses plus over refraction);
* Manifest astigmatism less than or equal to -1.00D;
* Soft contact lens wear in both eyes at least 5 days per week and at least 8 hours per day;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pregnant or lactating;
* Eye injury or surgery within twelve weeks immediately prior to enrollment;
* Any ocular condition that contraindicates contact lens wear;
* History of herpetic keratitis;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, including any use of topical ocular medications that would require instillation during contact lens wear, except for approved lubricating drops;
* Clinical significant dry eye not responding to treatment;
* Previous corneal or refractive surgery or irregular cornea;
* Requires reading glasses;
* Participation in a clinical trial (including contact lens or contact lens care product) within the previous 30 days;
* Wears habitual lenses in an extended wear modality (routinely sleeps in lenses overnight for 1 night per week or more) over the last 3 months prior to enrollment;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Nick, Dipl. Ing., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 study centers located in the US and 2 study centers located in Germany.
Pre-assignment Details: Of the 19 enrolled, 4 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants (15).
Groups:
- DAILIES TOTAL1/TRUEYE: Delefilcon A and narafilcon A contact lenses (1 in each eye) worn in a daily wear, daily disposable mode approximately 8 hours a day for approximately 1 week.
Period: Overall Study
Arm/Group | DAILIES TOTAL1/TRUEYE
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: This analysis group includes all randomized participants.
Arm/Group | DAILIES TOTAL1/TRUEYE
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Central Corneal Curvature From Dispense at Week 1
Description: Corneal curvature (horizontal and vertical keratometry values on the same eye) was measured using a calibrated keratometer prior to study lens dispense (Day 1) and approximately 15 minutes after study lens removal following 8 hours of wear (Week 1). Minus values in change-from-baseline indicate corneal flattening.
Time Frame: Dispense (Day 1 of lens wear), Week 1 (Day 8 of lens wear)
Population: This analysis group includes all randomized participants with data present at visit.
Measure: Mean (Standard Deviation); unit: diopters
Groups:
- DAILIES TOTAL1: Delefilcon A contact lens worn in 1 eye approximately 8 hours a day for 1 week
- TRUEYE: Narafilcon A contact lens worn in 1 eye approximately 8 hours a day for 1 week.
Arm/Group | DAILIES TOTAL1 | TRUEYE
Number analyzed (Participants) | 14 | 14
diopters | -0.44 (0.46) | -0.11 (0.26)

2. Secondary Outcome: Number of Eyes With Change of >1.00 Diopter (D) in Spherical Equivalent of Subjective Refraction From Baseline at Week 1
Description: Subjective manifest refraction was assessed using a phoropter or trial frame set with the subject's current prescription at Baseline (Visit 2) after a 2-day washout period and approximately 15 minutes after study lens removal following 8 hours of wear (Week 1). Spectacle over-refraction, if required, was performed. Higher myopia is indicated by larger negative values in manifest refraction.
Time Frame: Baseline, Week 1 (Day 8 of lens wear)
Population: This analysis group includes all randomized participants with data present at visit.
Measure: Number; unit: Eyes
Arm/Group | DAILIES TOTAL1 | TRUEYE
Number analyzed (Participants) | 14 | 14
Eyes | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (March, 2014 - May, 2014). This analysis group includes all participants/eyes exposed to the study products. Trial-fit lenses were not considered study products.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device.
Arm/Group | DAILIES TOTAL1 | TRUEYE
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DAILIES TOTAL1 (N=15) | TRUEYE (N=15)
Foreign body sensation in eyes (Eye disorders) | 1 | 0
Metamorphopsia (Eye disorders) | 1 | 1
Myokymia (Musculoskeletal and connective tissue disorders) | 1 | 1
Ocular discomfort (Eye disorders) | 1 | 0
Punctate keratitis (Eye disorders) | 1 | 0
Topography corneal abnormal (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.